CLINICAL TRIAL: NCT04255524
Title: OCTA to Quantify the Parapapillary Choroidal Microvascular Changes in High Myopia
Brief Title: Choroidal Change on OCTA in Eyes With High Myopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OCTAPPA
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Myopia, Progressive; Choroid Disease
Keywords: OCTA; Myopia; Choroid
MeSH Terms: conditions — Myopia, Degenerative; Choroid Diseases; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1/Control (Experimental): Spherical equivalent: -2.00～+2.00 D
  Interventions: Device: Optic coherence tomography angiography (OCTA)
- Group 1/Myopia (Experimental): Spherical equivalent: -3.00～-6.00 D
  Interventions: Device: Optic coherence tomography angiography (OCTA)
- Group 3/High (Experimental): Spherical equivalent: -6.00～-10.00 D
  Interventions: Device: Optic coherence tomography angiography (OCTA)
- Group 4/Super High (Experimental): Spherical equivalent: <-10.00
  Interventions: Device: Optic coherence tomography angiography (OCTA)

INTERVENTIONS:
Device: Optic coherence tomography angiography (OCTA) — Using non-invasive, repeatable, mature device OCTA to obtain choroidal angio-map

SUMMARY:
Myopia is a global healthy concern, especially the high myopia and pathological myopia among Asian populations. However, its mechanism still remains largely unclear. Recent findings suggested choroidal changes might be related to the development of myopia. This study is to useOCT angiography (OCT-A) to investigate parapapillary choroidal microvasculature change in myopic eyes, and try to find the cause-and-effect relationship between choroidal change and the development of myopia.

ELIGIBILITY:
Inclusion Criteria:

1. Spherical equivalent measurement can be included in above 4 groups
2. Willing to be followed up in the future 10 years

Exclusion Criteria:

1. Deny to sign the patient consent, or deny to be followed
2. Evidence of cardiac, or diabetic, or CNS disease.
3. Clinically diagnosed with retinal or choroidal disease
4. Glucoma
5. Cataract or corneal disease that influence the quality of fundus OCTA image

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Parapapillary choroidal microvasculature void (MvV) area | changes of MvV area from at 10 years
  area of parapapillary choroidal microvasculature void on OCTA images
Parapapillary choroidal microvasculature void (MvV) area | difference of MvV area in each group at baseline
  area of parapapillary choroidal microvasculature void on OCTA images
Parapapillary choroidal microvasculature void (MvV) area | changes of MvV area at 1 years
  area of parapapillary choroidal microvasculature void on OCTA images
Parapapillary choroidal microvasculature void (MvV) area | changes of MvV area at 3 years
  area of parapapillary choroidal microvasculature void on OCTA images
Parapapillary choroidal microvasculature void (MvV) area | changes of MvV area at 5 years
  area of parapapillary choroidal microvasculature void on OCTA images

SECONDARY OUTCOMES:
MvV number | baseline
  number of choroidal MvV with certain size
Correlation coefficient between choroidal MvV and refractive power | baseline
  Correlation coefficient between choroidal MvV and refractive power
Correlation coefficient between choroidal MvV and PPA area | baseline
  Correlation coefficient between choroidal MvV and parapapillary atrophy beta area
Correlation coefficient between choroidal MvV and choroid thickness | baseline
  Correlation coefficient between choroidal MvV and choroid thickness
Correlation coefficient between choroidal MvV and RNFL thickness | baseline
  Correlation coefficient between choroidal MvV and RNFL thickness
Correlation coefficient between choroidal MvV and Axial length | baseline
  Correlation coefficient between choroidal MvV and Axial length
Correlation coefficient between choroidal MvV and retinal parapapillary perfusion | baseline
  Correlation coefficient between choroidal MvV and retinal parapapillary perfusion on OCTA images.
Correlation coefficient between choroidal MvV and Macular perfusion | baseline
  Correlation coefficient between choroidal MvV and Macular perfusion on OCTA images, Retinal parapapillary perfusion with OCTA.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
After completion of the prospective observational study, we would like to share data for reasonable request from other researchers.